CLINICAL TRIAL: NCT03015194
Title: NHLBI DIR LAMPOON Study: Intentional Laceration of the Anterior Mitral Leaflet to Prevent Left Ventricular Outflow Tract Obstruction During Transcatheter Mitral Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999917032; 17-H-N032
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-03

CONDITIONS: Mitral Valve Failure
Keywords: LVOT (left ventricular outflow tract, obstruction); Transcatheter Mitral Valve Implantation; Transcatheter Heart Valve; Mitral Valve Regurgitation; Mitral Valve Stenosis
MeSH Terms: conditions — Bites and Stings; Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option (Experimental): The LAMPOON procedure has three steps: (1) leaflet traversal with a guidewire, followed by (2) leaflet laceration, immediately followed by (3) TMVR. These are all guided by fluoroscopy combined with transesophageal echocardiogram (TEE) or intracardiac echocardiography.
  Interventions: Device: Edwards SAPIEN 3 transcatheter heart valve; Device: ASHI INTECC Astato XS 20

INTERVENTIONS:
Device: Edwards SAPIEN 3 transcatheter heart valve — Used to relieve aortic stenosis in patients with symptomatic heart disease
  In this study it is not used for aortic stenosis-----the device is used in the mitral valve position.
Device: ASHI INTECC Astato XS 20 — The Astato 0.014" guidewire is used for transcatheter electrosurgery in two steps in this procedure. First it is used for leaflet traversal during electrification. This procedure is similar to the use of the Astato XS20 and an amputated Asahi Confienza Pro 12 in the transcaval IDE investigation recently published. Second, the midshaft is focally denuded and electrified for the leaflet traversal step.

SUMMARY:
Background:

Transcatheter mitral valve replacement (TMVR) is recommended for some people with mitral valve heart problems. But the usual TMVR techniques might cause an obstruction for some people. A new technique is called LAMPOON. It may have less risk of obstruction. Participants in this study will be among the first in the world to have this technique done.

Objectives:

To test the safety and effectiveness of the LAMPOON technique in TMVR.

Eligibility:

Adults ages 21 and over who are recommended to have TMVR with LAMPOON

Design:

Participants will be screened with medical history and exam and by review of medical records.

Participants will have blood tests, an ECG, a heart CT scan, and an echocardiogram before the procedure.

Participants will have TMVR with LAMPOON. They will have anesthesia or moderate sedation for the procedure. Doctors will use a wire to split the diseased mitral valve and move it out of the way before inserting the artificial mitral valve.

Participants will recover in an inpatient recovery unit.

They will repeat the previous tests before leaving the hospital, 1 month later, 6 months later and 1 year later. They will have yearly follow-up phone calls for about 5 years.

In the event of a participant's death, researchers will ask for an autopsy and to analyze the heart. Permission for this is not required as part of the study.

DETAILED DESCRIPTION:
Transcatheter mitral valve replacement (TMVR) is an option to treat mitral valve failure when no surgical options exist. In as many as half of patients, TMVR can cause life-threatening blockage of the left ventricle by displacing the existing mitral valve leaflet. For these patients the only options appear to avoid TMVR or in some to cause a focused heart attack and to wait 6 weeks. The investigators have developed and tested a technique to split the existing mitral valve leaflet and enable TMVR in patients who have no other options. The procedure is called intentional laceration of the anterior mitral leaflet to prevent left ventricular outflow tract obstruction (LAMPOON). Although there are no dedicated TMVR devices commercially available, there has been short-term success with implanted transcatheter aortic valve devices in the mitral position for TMVR.

The purpose of this study is to perform LAMPOON and TMVR in patients who have no good options to treat their mitral valve failure, using heart valve devices designed to implant in the aortic valve position.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adults age greater than or equal to 21 years
* Severe symptomatic native mitral valve failure after mitral annuloplasty repair or related to mitral annular calcification.
* Unacceptably high or prohibitive risk for surgical mitral valve replacement and indicated for transcatheter mitral valve replacement (TMVR) as determined by the multidisciplinary institutional heart team, including at least one cardiovascular surgeon who has examined the patient.
* High or prohibitive risk of LVOT obstruction (predicted neo-LVOT less than 200 mm2) or transcatheter heart valve dysfunction from long/redundant anterior mitral valve leaflet, as determined by the multidisciplinary institutional heart team.
* Anatomic eligibility for LAMPOON based on core lab assessment of the baseline CT and echocardiogram.
* Concordance of the study selection team

EXCLUSION CRITERIA

* Subjects unable to consent to participate, unless the subject has a legally authorized representative
* Subjects unwilling to participate or unwilling to return for study follow-up activities.
* Predicted neo-LVOT created by the Sapien-3 skirt, after LAMPOON, less than 150 mm2
* TAVR within 6 weeks
* Intended concurrent structural heart procedure, such as aortic or tricuspid valve implantation
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (6):
- United States (6):
  - Medstar Washington Hospital Center, Cardiovascular Research Program, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - University of Washington Division of Cardiology, Seattle, Washington

REFERENCES:
- [Derived] Khan JM, Babaliaros VC, Greenbaum AB, McCabe JM, Rogers T, Eng MH, Foerst JR, Yazdani S, Paone G, Gleason PT, Halaby RN, Bruce CG, Tian X, Stine AM, Lederman RJ. 5-Year Outcomes of Anterior Mitral Leaflet Laceration to Prevent Outflow Obstruction. JACC Cardiovasc Interv. 2024 Sep 23;17(18):2157-2167. doi: 10.1016/j.jcin.2024.05.041. Epub 2024 Sep 4. PMID 39243268
- [Derived] Khan JM, Babaliaros VC, Greenbaum AB, Foerst JR, Yazdani S, McCabe JM, Paone G, Eng MH, Leshnower BG, Gleason PT, Chen MY, Wang DD, Tian X, Stine AM, Rogers T, Lederman RJ. Anterior Leaflet Laceration to Prevent Ventricular Outflow Tract Obstruction During Transcatheter Mitral Valve Replacement. J Am Coll Cardiol. 2019 May 28;73(20):2521-2534. doi: 10.1016/j.jacc.2019.02.076. PMID 31118146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol enrolled 32 participants, however 2 participants had screen failed.
Groups:
- Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option: The intentional laceration of the anterior mitral leaflet to prevent left ventricular outflow tract obstruction (LAMPOON) is a one-time procedure on Day 0 with three steps: (1) leaflet traversal with a guidewire, followed by (2) leaflet laceration, immediately followed by (3) TMVR. These are all guided by fluoroscopy combined with transesophageal echocardiogram (TEE) or intracardiac echocardiography.
Period: Overall Study
Arm/Group | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option
Started | 30
Completed | 18
Not Completed | 12
Not completed — Death | 10
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 76 [47 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With "Acceptable" Technical Success of the LAMPOON Procedure
Description: Participants post intentional laceration of the anterior mitral leaflet to prevent left ventricular outflow tract obstruction (LAMPOON) procedure that were defined as an "acceptable technical success" met the following criteria:
  * Successful LAMPOON traversal and laceration; and
  * Peak LVOT gradient < 50 mm Hg; and
  * Absence of procedural mortality; and
  * Successful access, delivery, and retrieval of the LAMPOON device system; and
  * Successful deployment and correct positioning of the first intended device; and
  * Freedom from emergency surgery or reintervention related to the device or access procedure.
  The first two factors are modifications of the MVARC (mitral valve academic research consortium) consensus endpoint, specific for LAMPOON procedure.
Time Frame: Exit from the Cardiac Catheterization Laboratory
Measure: Number; unit: participants
Groups:
- Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option: The intentional laceration of the anterior mitral leaflet to prevent left ventricular outflow tract obstruction (LAMPOON) is a one-time procedure on Day 0 with three steps: (1) leaflet traversal with a guidewire, followed by (2) leaflet laceration, immediately followed by (3) TMVR. These are all guided by fluoroscopy combined with transesophageal echocardiogram (TEE)or intracardiac echocardiography.
Arm/Group | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option
Number analyzed (Participants) | 30
participants
  Successful LAMPOON traversal and laceration | 30
  LVOT gradient <50 mm Hg | 30
  Procedure survival | 30
  Successful access, delivery, and retrieval of LAMPOON device system | 30
  Successful deployment and correct positioning of the first intended device | 27
  Freedom from emergency surgery or reintervention related to the device or access procedure | 22

2. Primary Outcome: Number of Participants With "Optimal" Technical Success of the LAMPOON Procedure
Description: Participants post intentional laceration of the anterior mitral leaflet to prevent left ventricular outflow tract obstruction (LAMPOON) procedure that were defined as an "acceptable technical success" met the following criteria:
  * Successful LAMPOON traversal and laceration; and
  * Peak LVOT gradient < 30 mm Hg; and
  * Absence of procedural mortality; and
  * Successful access, delivery, and retrieval of the LAMPOON device system; and
  * Successful deployment and correct positioning of the first intended device; and
  * Freedom from emergency surgery or reintervention related to the device or access procedure.
  The first two factors are modifications of the MVARC (mitral valve academic research consortium) consensus endpoint, specific for LAMPOON procedure.
Time Frame: Exit from the Cardiac Catheterization Laboratory
Measure: Number; unit: participants
Arm/Group | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option
Number analyzed (Participants) | 30
participants
  Successful LAMPOON traversal and laceration | 30
  LVOT gradient <30 mm Hg | 29
  Procedure survival | 30
  Successful access, delivery, and retrieval of LAMPOON device system | 30
  Successful deployment and correct positioning of the first intended device | 30
  Freedom from emergency surgery or reintervention related to the device or access procedure | 22

ADVERSE EVENTS:
Time Frame: Adverse event recording will start on Day (0) until 30-day follow up, after this only serious adverse events (SAE), serious adverse device effects (SADE), unanticipated device effects (UADE) and unanticipated problems (UP) will be reported to the Sponsor for 1 year.
Arm/Group | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option
All-Cause Mortality (participants affected / at risk) | 16/30
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option (N=30)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 10 (20)
Arterial injury (Injury, poisoning and procedural complications) | 3 (4)
Atrioventricular Block complete (Cardiac disorders) | 2 (2)
Bacteremia (Infections and infestations) | 2 (4)
Cardiac arrest (Cardiac disorders) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Perivalvular leak (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 5 (5)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac disorders other-LVOT obstruction post TMVR. (Cardiac disorders) | 1 (1)
Cardiac disorders-other -increased mitral valve gradient, TMVR thrombus (Cardiac disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Cardiac disorders-other-left apical pseudoaneurism. (Cardiac disorders) | 1 (1)
Cardiac disorders-other-increased LVOT gradient post TMVR (Cardiac disorders) | 2 (2)
Cardiac disorders-other-elevated mitral valve gradient ; possible TMVR thrombus (Cardiac disorders) | 1 (1)
Cardiac disorders-other-perivalvular leak post TMVR (Cardiac disorders) | 2 (2)
Cardiac disorders-other-perivalvular pseudoaneurysm. (Cardiac disorders) | 1 (1)
Cardiac disorders-other-mitral valve thrombus (Cardiac disorders) | 1 (1)
tenting of anterior leaflet of mitral valve causing myocardial dysfunction and severe hypotension (Cardiac disorders) | 1 (1)
Cardiac disorders-other-severe perivalvular leak immediately post TMVR (Cardiac disorders) | 1 (1)
Cardiac disorders-other-right ventricular apex pseudoaneurysm (Cardiac disorders) | 1 (1)
chest pain-cardiac (Cardiac disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
endocarditis infective (Infections and infestations) | 1 (1)
endocarditis infective (Cardiac disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (2)
fall (Injury, poisoning and procedural complications) | 3 (4)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 3 (3)
Gastrointestional disorders -other-Toxic Megacolon (Gastrointestinal disorders) | 1 (1)
Gastrointestional disorders -other-cholecystitis (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions-other-AV fistual bleed. (General disorders) | 1 (1)
General disorders and administration site conditions-other-AV fistual thrombosed. (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 9 (16)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 9 (12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations-other-C. Difficile infection (Infections and infestations) | 1 (1)
Infections and infestations-other-septic emboli (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications-other-digoxin toxicity (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications-other-Coumadin toxicity (Injury, poisoning and procedural complications) | 3 (3)
Injury, poisoning, and procedureal complications-other-opioid toxicity (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications-other-subtherapeutic INR-coumadin (Injury, poisoning and procedural complications) | 1 (1)
Investigations other-guidewire fracture and separation (Investigations) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Investigations other-TMVR embolized (Investigations) | 1 (1)
Investigations other-TMVR dehiscence (Investigations) | 1 (1)
Investigations-other-explant of TMVR Sapien -3 due to malpositioning, MAC, and LV calcification (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 (5)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Musculoskeletal and connective tissue disorder-other-generalized pain with impending death (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
pain (General disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (3)
Respiratory , thoracic and mediastinal disorders-other-pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory , thoracic and mediastinal disorders-other-pneumonia with sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory, thoracic and mediastinal disorders-other-COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders-other-excessive secretions while intubated. (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 4 (7)
Stroke (Nervous system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Surgical and Medical Procedures-others-alcohol septal ablation to treat LVOT obstruction (Surgical and medical procedures) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular disorder-other-thrombolic event (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vascular disorders-other-hypotensive shock post cardiac arrest (Vascular disorders) | 1 (1)
vascular disorders-other-thrombotic event (Vascular disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (3)
Ventricular Tachycardia (Cardiac disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laceration of Anterior Mitral Leaflet in Mitral Valve Failure Participants With no Surgical Option (N=30)
Acidosis (Metabolism and nutrition disorders) | 4 (5)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 28 (32)
Anxiety (Psychiatric disorders) | 5 (7)
Arterial thromboembolism (Vascular disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 5 (6)
Atrioventricular block first degree (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder Infection (Infections and infestations) | 2 (2)
Blood and Lymphatic systems disorder, other-Elevated WBCs (Blood and lymphatic system disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 5 (5)
Blood lactate dehydrogenase increased (Investigations) | 7 (7)
Cardiac disorders other-LVOT obstruction (Cardiac disorders) | 2 (2)
Cardiac disorders other-TMVR perivalvular link (Cardiac disorders) | 5 (6)
Cardiac troponin I increase (Investigations) | 27 (30)
Chest pain - cardiac (Cardiac disorders) | 4 (10)
conduction disorder (Cardiac disorders) | 5 (6)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Reproductive system and breast disorders) | 5 (6)
Creatinine increased (Investigations) | 15 (19)
Delirium (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
dysphagia (Gastrointestinal disorders) | 3 (3)
Edema Limbs (General disorders) | 6 (6)
Ejection fraction decreased (Investigations) | 10 (10)
Encephalopathy (Nervous system disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fever (General disorders) | 3 (3)
General disorders and administration sites, other-AV fistual bleed (General disorders) | 2 (4)
Haptoglobin decrease (Investigations) | 4 (4)
headache (Nervous system disorders) | 2 (2)
Heart failure (Cardiac disorders) | 24 (36)
hematoma (Vascular disorders) | 10 (11)
hematuria (Renal and urinary disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 12 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 12 (14)
INR increased (Investigations) | 12 (17)
Investigations other-albumin low (Investigations) | 3 (4)
Investigations other-decreased INR (Investigations) | 6 (9)
Investigations, other-Calcium decreased (Investigations) | 5 (5)
Investigations other-sodium low (Investigations) | 6 (7)
Investigations other-low magnesium (Investigations) | 2 (2)
Investigations other-potassium high (Investigations) | 3 (5)
Investigations other-potassium low (Investigations) | 6 (8)
Leukocytosis (Blood and lymphatic system disorders) | 16 (20)
Lower gastrointestional hemorrhage (Gastrointestinal disorders) | 3 (3)
Malaise (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 4 (4)
Platelet Count Decrease (Investigations) | 28 (34)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders, other-pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediatinal disorders other-Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediatinal disorders other-Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
thromboembolic event (Vascular disorders) | 2 (2)
Upper gastrointestional hemorrhage (Gastrointestinal disorders) | 3 (3)
urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infections (Infections and infestations) | 6 (6)
vascular disorders other-bruise (Vascular disorders) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Wound Infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03015194/Prot_SAP_000.pdf